CLINICAL TRIAL: NCT03029117
Title: Prospective Cohort Study Compares Effect of Corrected and Uncorrected Rheumatic Heart Valve of Pregnant Women on Maternal and Fetal Outcomes
Brief Title: Effect of Rheumatic Heart Disease on Maternal and Fetal Outcomes
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Armia Michael, resident physician, Assiut University
Other Study IDs: 12345
Record Dates: First submitted 2017-01-19; First posted 2017-01-24 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Rheumatic; Heart Disease, Maternal, Affecting Fetus
Keywords: rheumatic pregnancy
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- corrected and uncorrected rheumatic valve lesions
  Interventions: Procedure: correction of rheumatic valve lesions

INTERVENTIONS:
Procedure: correction of rheumatic valve lesions

SUMMARY:
It's prospective Cohort study to compare maternal and fetal outcomes in pregnant females between corrected and uncorrected rheumatic valve lesions

DETAILED DESCRIPTION:
Heart disease is one of the most important medical complications during pregnancy as it is one of the common, indirect obstetric causes of maternal death. Approximately 1% of pregnancies are complicated by cardiac disease .

Rheumatic heart disease (RHD) is the most common acquired heart disease in pregnancy RHD is a chronic acquired heart disorder resulting from acute rheumatic fever. In developing countries, RHD continues to be a major cause of cardiac morbidity and mortality especially among young adult females In pregnancies complicated with cardiac disorders, maternal and perinatal mortality and morbidity depend on the type of disorder, the functional status of the patient and the complications associated with the pregnancy.

Mitral stenosis is the most common valvular lesion in women with rheumatic heart disease, remains the most common acquired valvular lesion in pregnant women and the most common cause of maternal death from cardiac causes .

Although mortality is not high in women, the rate of fetal morbidity rises with the severity of mitral stenosis from 14% in pregnant patients with mild mitral stenosis , to 28% in women with moderate mitral stenosis and 33% in pregnant patients with severe mitral stenosis (area <1.5 CM2).

In the second and third trimesters, when maternal blood volume and cardiac output peak, heart failure may occur in pregnant women with moderate or severe mitral stenosis, even in previously asymptomatic women .

The rates of prematurity in fetus of women with rheumatic heart diseases are 20% to 30%, fetal growth restriction 5% to 20%, and stillbirth (1% to 3%).

The advancement in cardiology and obstetrics has provided major improvements in the management of pregnant patients with cardiac disorders. Now we are facing more women with previous history of surgical correction of rheumatic heart disease.

Vaginal delivery is considered In women with mild mitral stenosis, and in patients with moderate mitral stenosis ,. Even in women with severe MS in whom symptoms are New York Heart Association (NYHA) Class I-II without pulmonary hypertension, vaginal delivery is considered Cesarean section may be preferred in patients with severe mitral stenosis with NYHA Class III-IV symptoms, or who have pulmonary hypertension despite medical therapy.

Therapeutic options for in women with rheumatic heart disease include both medical and surgical alternatives, as well as catheter-based interventions The choice dependent on the degree of valvular affection and patient symptoms. There are few studies that compare the Maternal and fetal outcomes in women with rheumatic heart disease between patient with corrected and uncorrected valve lesions

ELIGIBILITY:
Inclusion Criteria:

* pregnant females with rheumatic heart disease

Exclusion Criteria:

* other heart diseases ( cardiomyopathy , myocardial infarction ...etc.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: pregnant females with rheumatic heart disease come for antenatal care at out patient clinic at tertiary obstetric center
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
maternal morbidity | 40 days after delivery
  compare maternal morbidity between corrected and uncorrected valve lesions in pregnant women

SECONDARY OUTCOMES:
Fetal outcome | first 1 day after delivery
  compare birth weight and need for admission at neonatal intensive care unit (NICU) between corrected and uncorrected valve lesions in pregnant women

IPD SHARING:
Plan to Share IPD: No